CLINICAL TRIAL: NCT00537446
Title: Effect of Noninvasive Positive Pressure Ventilation on Pulmonary Function Testing in Amyotrophic Lateral Sclerosis
Brief Title: Effect of Noninvasive Ventilation on Lung Function in Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Robert C. Basner, Special Lecturer in Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAC7394
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: noninvasive ventilation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-level ventilation (Active Comparator): Each subject will spend 2 hours receiving high-level noninvasive ventilation.
  Interventions: Device: noninvasive positive pressure ventilation
- Low-level ventilation (Active Comparator): Each subject will receive 2 hours of low-level noninvasive positive pressure ventilation.
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive positive pressure ventilation — Each subject will undergo 2 hours of high-level noninvasive positive pressure ventilation, with an inspiratory positive airway pressure of 12 cm H2O and an expiratory positive airway pressure of 3 cm H2O.
  Other Names: "BiPAP" (Respironics), variable positive airway pressure (VPAP) (ResMed), bilevel positive airway pressure, noninvasive ventilation
  Arms: High-level ventilation
Device: noninvasive positive pressure ventilation — Each subject will undergo 2 hours of low-level noninvasive positive pressure ventilation, with an inspiratory positive airway pressure of 6 cm H2O and an expiratory positive airway pressure of 3 cm H2O.
  Other Names: BiPAP (Respironics), VPAP (ResMed), bilevel positive airway pressure, noninvasive ventilation
  Arms: Low-level ventilation

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS), or "Lou Gehrig's Disease", is a fatal disorder that causes progressive degeneration and weakening of the muscles of breathing, leading to breathing insufficiency and eventually breathing failure. This breathing insufficiency is commonly treated with a breathing assistance device, known as noninvasive positive pressure ventilation (NIPPV). While generally well tolerated and accepted, it is not clear whether or to what extent NIPPV in fact helps breathing function: some data suggest that NIPPV preserves breathing function over time, whereas other data suggest that it actually causes breathing function to decline more quickly. No studies have shown what the acute effect of NIPPV is on breathing muscle function in ALS patients.

This study will test the hypothesis that the acute use of NIPPV, at pressure levels that are in common clinical use, will cause measurable changes in tests of breathing function, compared to baseline and to lower levels of NIPPV. We expect that the results of this study will help to clarify whether and to what extent NIPPV assists respiratory muscle function in patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of amyotrophic lateral sclerosis
* clinical indication to start noninvasive ventilation (forced vital capacity < 50% predicted or signs/symptoms of respiratory insufficiency)
* age 18 to 80 years old

Exclusion Criteria:

* prior institution of NIPPV
* inability to safely use NIPPV
* indications for tracheostomy assisted ventilation because of inability to clear secretions from the airway
* inability or unwillingness to perform pulmonary function testing
* presence of advanced dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Basner, MD, Principal Investigator — Columbia University
Locations (1):
- Eleanor and Lou Gehrig ALS/MDA Center at Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Level and Low Level Ventilation: All participants are listed as one group, as the breakdown per Arm/Group is not available (PI no longer has raw data on file).
Period: Overall Study
Arm/Group | High Level and Low Level Ventilation
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- High Level and Low Level Ventilation: All participants
Arm/Group | High Level and Low Level Ventilation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pulmonary Function and Respiratory Muscle Pressure Testing
Time Frame: 5 hours
Population: Data were collected but not analyzed as specified in the title because the sample size does not generate enough statistical significance. PI no longer has raw data on file. All efforts have been made to retrieve the data and data could not be recovered.
Arm/Group | High-level Ventilation | Low-level Ventilation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Difference in Gas Exchange
Time Frame: 5 hours
Population: as for outcome 1
Arm/Group | High-level Ventilation | Low-level Ventilation
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Difference in Subjective Dyspnea Between Baseline and the Two Different Ventilator Modes
Time Frame: 5 hours
Population: as for outcome 1
Arm/Group | High-level Ventilation | Low-level Ventilation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 hours
Description: No adverse events were observed.
Arm/Group | High-level Ventilation | Low-level Ventilation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes